CLINICAL TRIAL: NCT05784493
Title: The Effect of Intraabdominal Saline Washing After Laparoscopic Hysterectomy on Postoperative Pain: Double Blind Randomized Controlled Study
Brief Title: Pain After Laparoscopic Hysterectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Namik Kemal University (Other)
Collaborators: Fırat Can Sogut (Unknown); Ozlem Sevinc Ergul (Unknown); Mehmet Veysel Arın (Unknown)
Responsible Party: Principal Investigator, Mehmet Baki Senturk, Pirincipal İnvestigator, Namik Kemal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2020.04.06.02
Record Dates: First submitted 2023-03-02; First posted 2023-03-27 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Washing by heated saline group (Experimental)
  Interventions: Other: Study group
- Washing by normal room temperature saline group (Active Comparator)
  Interventions: Other: Study group

INTERVENTIONS:
Other: Study group — Washing by heated saline group

SUMMARY:
The investigators evaluated postoperative pain after total laparoscopic hysterectomy. Two arm are evaluated. During laparoscopic hysterectomy, in one arm; abdominal cavity was washed by saline at normal room temperature. In another arm; abdominal cavity was washed heated saline . Postoperative pain was evaluated by using visual analogy scale.

DETAILED DESCRIPTION:
The aim of this study was evaluated the effect of washing abdominal cavity by heated or normal temperature saline on postoperative pain.

This study is double blind randomized controlled study.

inclusion criteria: all of cases that had laparoscopic hysterectomy for bening condition

exclusion criteria: maling cases and conversion to laparotomy

after randomization and completion of surgery, investigator was evaluated postoperative pain at 0-4-8 th hours by using visual analog scale participants and investigator were blinded .

ELIGIBILITY:
Inclusion Criteria:

* all of cases that had laparoscopic hysterectomy for bening conditions

Exclusion Criteria:

* maling cases
* conversion to laparotomy

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Pain assessed by visual analog scale | 5 months
  To assess postoperative pain incidence by using visual analog scale

CONTACTS AND LOCATIONS:
Locations (1):
- Namik Kemal University, Tekirdağ, Turkey (Türkiye)